CLINICAL TRIAL: NCT06935526
Title: The Effect of a Mobile Education Program and Telephone Monitoring Developed for Patients With Implantable Cardioverter Defibrillators on Shock Anxiety, Device Acceptance, and Self-Efficacy
Brief Title: Mobile Education and Telephone Monitoring for ICD Patients: Effects on Anxiety, Acceptance, and Self-Efficacy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Mediha SERT, Principal Investigator, research assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 527; 2024.7 (Other Grant/Funding Number: VEHBİ KOÇ FOUNDATION NURSING FUND)
Record Dates: First submitted 2025-03-24; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Patient Acceptance of Health Care; Nursing; Implantable Cardioverter Defibrillator (ICD); Self-Efficacy; Shock, Cardiogenic
Keywords: Device acceptance; shock anxiety; implantable cardioverter defibrillator; self-efficacy; nursing
MeSH Terms: conditions — Patient Acceptance of Health Care; Shock, Cardiogenic

STUDY DESIGN:
Who Masked: Participant
Masking Description: All patients were administered a mobile education program, and the groups to which the patients belonged were not disclosed, ensuring that the patients were blinded. The aim was to achieve single blinding by ensuring that participants were unaware of which group they were assigned to. Additionally, it was planned to minimize bias by not providing information to the person conducting the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group of mobile education programe (Experimental): The intervention group consists of 44 patients attending routine ICD follow-ups. Patients completed a pre-test before the intervention and a post-test at 12 weeks via M-ICDEP. Data were collected using FSAS, FPAS, OE-ICD, and SB-ICD scales on M-ICDEP. A shock management simulation was conducted at both pre-and post-tests, evaluated with the Shock Management Control Form, and added to shock anxiety data.
  The intervention group used M-ICDEP anytime during the 3-month follow-up, which includes three sections: education, summary information, and shock management simulation. The program aimed to reduce shock-related anxiety, increase device acceptance, and enhance self-efficacy. Telephone follow-ups were conducted in the 2nd, 5th, and 8th weeks, evaluating patients using the Telephone Calls Monitoring Form. The information shared during these calls was continued within the training program's scope, ensuring consistent reinforcement of the content.
  Interventions: Other: The mobile training program and telephone follow-ups
- Standard Treatment Group (Active Comparator): The control group consists of 44 patients attending routine ICD follow-ups. Patients completed a pre-test before the intervention and a post-test at 12 weeks via M-ICDEP. Data were collected using FSAS, FPAS, OE-ICD, and SB-ICD scales on M-ICDEP. A shock management simulation was conducted at both pre-and post-tests, evaluated with the Shock Management Control Form, and added to shock anxiety data. The control group used M-ICDEP, which includes only one section: summary information, anytime during the 3-month follow-up. The program aimed to reduce shock-related anxiety, increase device acceptance, and enhance self-efficacy. Routine outpatient follow-up was continued for the control group without any other intervention.
  Interventions: Other: Only a two-page summary section of M-ICDEP

INTERVENTIONS:
Other: The mobile training program and telephone follow-ups — The study had three phases: pre-test, implementation, and post-test. Data were collected twice, before the intervention and in the third month, using validated scales and a shock management simulation via the mobile training program (M-ICDEP). M-ICDEP included three sections: an educational section, a two-page summary, and a shock management simulation. All sections were shared with the intervention group. After the pre-test, intervention group patients could log in to M-ICDEP anytime using their email and password, accessing content repeatedly during the three-month follow-up. The researcher conducted telephone follow-ups in the second, fifth, and eighth weeks, evaluating patients using the Telephone Calls Monitoring Form. The information given to the patients during the telephone conversation was continued within the limited of the training program prepared within the scope of M-ICDEP.
  Arms: The group of mobile education programe
Other: Only a two-page summary section of M-ICDEP — The study had three phases: pre-test, implementation, and post-test. Data were collected twice, before the intervention and in the third month, using validated scales and a shock management simulation via the mobile training program (M-ICDEP). M-ICDEP included three sections: an educational section, a two-page summary, and a shock management simulation. Only a two-page summary section were shared with the control group. After the pre-test, control group patients could log in to M-ICDEP anytime using their email and password, accessing the summary section repeatedly during the three-month follow-up. Routine outpatient follow-up was continued for the control group without any other intervention.
  Arms: Standard Treatment Group

SUMMARY:
Aim: This study was conducted to determine the effect of a mobile education program and telephone monitoring developed for patients with implantable cardioverter defibrillators (ICD) on shock anxiety, device acceptance, and self-efficacy.

Method: The study was designed as a single-blind, randomized controlled trial consisting of two phases. In the first phase, the Mobile ICD Education Program (M-ICDEP) was developed. In the second phase, the effectiveness of M-ICDEP was evaluated through a randomized controlled design with 88 ICD patients who attended routine battery check-ups.

Research data were collected through the mobile education program using the Personal Information Form, Florida Shock Anxiety Scale (FSAS), Florida Patient Acceptance Scale (FPAS), and the Self-Efficacy and Outcome Expectations Scales After ICD Implantation (OE-ICD and SB-ICD). Additionally, patients underwent a shock management simulation via M-ICDEP, and their data were assessed using the Shock Management Control Form, which was included in the evaluation of shock anxiety.

Patients in both the intervention and control groups used M-ICDEP for three months. The control group had access only to the brief educational booklet section containing general information, while the intervention group had access to all sections. Patients in the intervention group also received telephone follow-ups during the second, fifth, and eighth weeks of the monitoring period. Data were collected twice: once before the intervention (pre-test) and once in the third month (post-test). Statistical analyses will conducted using the SAS 9.4 software package.

DETAILED DESCRIPTION:
1. Definition and Importance of the Problem

   Implantable cardioverter defibrillators (ICDs) are devices developed to prevent sudden cardiac death resulting from ventricular arrhythmias. According to the 2017 guidelines of the European Heart Rhythm Association, the annual number of ICD implantations per million people is reported to be 107 worldwide and 115 in Turkey. Furthermore, over the past decade, implantation rates have increased by 44% globally and 804.1% in Turkey. Although ICD therapy has been proven to reduce mortality by 28-40% and is more effective than antiarrhythmic drugs, living with an ICD can lead to various psychosocial problems in patients. In particular, anxiety and device adaptation problems are frequently encountered after implantation.

   The foreign nature of the ICD, concerns about living dependently on the device, its activation during potentially fatal arrhythmias, and its capability to deliver shocks contribute to increased anxiety. Studies indicate that 44-55% of patients experience shock-related anxiety, with uncertainty regarding the sensation, location, and timing of shocks exacerbating this distress. Additionally, 95% of individuals who have experienced a shock develop anxiety. Anxiety and shock experiences can hinder device acceptance, adversely affecting patients' daily lives. It has been reported that individuals struggling with device acceptance exhibit lower levels of self-efficacy and that self-efficacy plays a crucial psychological role in disease adaptation. Consequently, assessing patients' self-efficacy is of significant importance.

   Adequate patient education, telephone follow-ups, and continuous care have been shown to enhance device acceptance and self-efficacy. Despite the recognized importance of patient education and follow-up, 97% of ICD patients report needing further education and monitoring, suggesting a gap in the provision of necessary training.

   Currently, innovative and interactive educational methods, such as mobile health applications and simulation techniques, are widely used for patient education. Mobile applications facilitate easy access to information, while simulation methods provide a realistic learning environment by allowing patients to experience real-life scenarios. While international literature includes studies on the use of mobile health applications for ICD patient monitoring, no studies have been identified that apply a mobile education program. Therefore, this study is expected to contribute innovatively to the literature by providing a realistic learning environment through a mobile education program incorporating different algorithms and a shock management simulation. Additionally, it is hypothesized that mobile education programs and telephone monitoring may improve patients' shock anxiety, device acceptance, and self-efficacy levels.

   ---
2. Aim of the Study

This study aims to determine the effect of a mobile education program and telephone monitoring developed for ICD patients on shock anxiety, device acceptance, and self-efficacy. It has been designed as a single-blind, randomized controlled trial consisting of two phases. The first phase involves the development of the mobile education program, while the second phase aims to evaluate the impact of the program on patients' shock anxiety, device acceptance, and self-efficacy.

* Research Hypotheses

The research hypotheses are formulated as follows:

Compared to the control group, ICD patients in the intervention group who receive the mobile education program and telephone monitoring will experience:

1. H1: A decrease in shock anxiety levels.
2. H1: An increase in device acceptance levels.
3. H1: An increase in self-efficacy and outcome expectations levels.

ELIGIBILITY:
Inclusion Criteria:

* Having an ICD implant
* Being able to read and write
* Being 18 years of age or older
* Not having a cognitive or communication disability
* Not having a diagnosed psychiatric disease
* Not having a generalized anxiety disorder (GAD-7 test score <8)*
* Not having a vision problem to the extent that it prevents the use of technological devices
* Having the knowledge and skills to use technological devices
* Having a smartphone that runs on the Android operating system and has internet access
* Agreeing to participate in the study

Exclusion Criteria:

* Patient not continuing after the second telephone follow-up phase of the study
* Not using the mobile application regularly (frequency of use monitored by the application)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Shock anxiety level | three month
  Shock anxiety is measured using the Florida Shock Anxiety Scale (FSAS), which includes 10 items. Scores range from 5 to 50. Higher scores indicate higher levels of shock-related anxiety.
The device acceptance levels | three month
  Device acceptance is evaluated with the Florida Patient Acceptance Scale (FPAS), which contains 18 items. The total score ranges from 15 to 75. Higher scores reflect greater acceptance of the implanted cardioverter defibrillator.
Self-efficacy and outcome expectation levels | three month
  Self-efficacy and outcome expectations are assessed using the Self-Efficacy and Outcome Expectations Scale, based on the ICD Internet Intervention model. It has two subscales: self-efficacy (16 items) and outcome expectations (7 items). The total score ranges from 7 to 195. Higher scores in both subscales indicate higher self-efficacy and more positive outcome expectations.

CONTACTS AND LOCATIONS:
Overall Officials: Mediha SERT GÖKÇEBEL, Researcher, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared; however, summary statistics (mean, standard deviation, frequencies, etc.) will be included in the thesis and relevant publications

REFERENCES:
- [Background] Zipes DP. First conclusive evidence that the implantable cardioverter-defibrillator reduces total mortality compared with drugs. Heart Rhythm. 2024 Jan;21(1):4-5. doi: 10.1016/j.hrthm.2023.09.025. No abstract available. PMID 38176770
- [Background] Wilson MH, Engelke MK, Sears SF, Swanson M, Neil JA. Disease-specific quality of life-patient acceptance: racial and gender differences in patients with implantable cardioverter defibrillators. J Cardiovasc Nurs. 2013 May-Jun;28(3):285-93. doi: 10.1097/JCN.0b013e31824e072e. PMID 22580627
- [Background] Tsuji Y, Heijman J, Nattel S, Dobrev D. Electrical storm: recent pathophysiological insights and therapeutic consequences. Basic Res Cardiol. 2013 Mar;108(2):336. doi: 10.1007/s00395-013-0336-2. Epub 2013 Feb 21. PMID 23429935
- [Background] Steiner JM, Bernacki G, Kirkpatrick J. My guardian angel: patients' fears and desires related to discussing implantable cardioverter-defibrillator deactivation. Heart. 2020 Feb;106(3):168-169. doi: 10.1136/heartjnl-2019-315935. Epub 2019 Oct 31. No abstract available. PMID 31672781
- [Background] Sportsman S, Schumacker RE, Hamilton P. Evaluating the impact of scenario-based high-fidelity patient simulation on academic metrics of student success. Nurs Educ Perspect. 2011 Jul-Aug;32(4):259-65. doi: 10.5480/1536-5026-32.4.259. PMID 21923008
- [Background] Sears SF, Matchett M, Conti JB. Effective management of ICD patient psychosocial issues and patient critical events. J Cardiovasc Electrophysiol. 2009 Nov;20(11):1297-304. doi: 10.1111/j.1540-8167.2009.01526.x. Epub 2009 Jun 26. PMID 19563356
- [Background] Pavia S, Wilkoff B. The management of surgical complications of pacemaker and implantable cardioverter-defibrillators. Curr Opin Cardiol. 2001 Jan;16(1):66-71. doi: 10.1097/00001573-200101000-00010. PMID 11124721
- [Background] Morken IM, Bru E, Norekval TM, Larsen AI, Idsoe T, Karlsen B. Perceived support from healthcare professionals, shock anxiety and post-traumatic stress in implantable cardioverter defibrillator recipients. J Clin Nurs. 2014 Feb;23(3-4):450-60. doi: 10.1111/jocn.12200. Epub 2013 Sep 17. PMID 24102743
- [Background] Mond HG, Proclemer A. The 11th world survey of cardiac pacing and implantable cardioverter-defibrillators: calendar year 2009--a World Society of Arrhythmia's project. Pacing Clin Electrophysiol. 2011 Aug;34(8):1013-27. doi: 10.1111/j.1540-8159.2011.03150.x. Epub 2011 Jun 27. PMID 21707667
- [Background] Mattsson G, Magnusson P. Long-term follow-up of implantable cardioverter defibrillator patients with regard to appropriate therapy, complications, and mortality. Pacing Clin Electrophysiol. 2020 Feb;43(2):245-253. doi: 10.1111/pace.13869. Epub 2020 Jan 22. PMID 31891421
- [Background] Marcus GM, Chan DW, Redberg RF. Recollection of pain due to inappropriate versus appropriate implantable cardioverter-defibrillator shocks. Pacing Clin Electrophysiol. 2011 Mar;34(3):348-53. doi: 10.1111/j.1540-8159.2010.02971.x. Epub 2010 Nov 15. PMID 21077915
- [Background] Lemon J, Edelman S, Kirkness A. Avoidance behaviors in patients with implantable cardioverter defibrillators. Heart Lung. 2004 May-Jun;33(3):176-82. doi: 10.1016/j.hrtlng.2004.02.005. PMID 15136777
- [Background] Kuhl EA, Dixit NK, Walker RL, Conti JB, Sears SF. Measurement of patient fears about implantable cardioverter defibrillator shock: an initial evaluation of the Florida Shock Anxiety Scale. Pacing Clin Electrophysiol. 2006 Jun;29(6):614-8. doi: 10.1111/j.1540-8159.2006.00408.x. PMID 16784427
- [Background] Khani SAG, Matourypour P, Haghjoo M, Zakerimoghadam M. The Effect of Continuous Care Program on the Self-Efficacy of Patients with Implantable Cardioverter Defibrillator: A Randomized Control Trial. Iran J Nurs Midwifery Res. 2023 Jul 24;28(4):455-460. doi: 10.4103/ijnmr.ijnmr_467_21. eCollection 2023 Jul-Aug. PMID 37694212
- [Background] Heidari M, Harandi PN, Moghaddasi J, Kheiri S, Azhari A. Effect of Home-Based Cardiac Rehabilitation Program on Self-Efficacy of Patients With Implantable Cardioverter Defibrillator. SAGE Open Nurs. 2023 Apr 24;9:23779608231166473. doi: 10.1177/23779608231166473. eCollection 2023 Jan-Dec. PMID 37124375
- [Background] Hacihasanoglu R, Gozum S, Capik C. Validity of the Turkish version of the medication adherence self-efficacy scale-short form in hypertensive patients. Anadolu Kardiyol Derg. 2012 May;12(3):241-8. doi: 10.5152/akd.2012.068. Epub 2012 Mar 2. PMID 22381924
- [Background] Glikson M, Friedman PA. The implantable cardioverter defibrillator. Lancet. 2001 Apr 7;357(9262):1107-17. doi: 10.1016/S0140-6736(00)04263-X. PMID 11297981
- [Background] Gehi AK, Mehta D, Gomes JA. Evaluation and management of patients after implantable cardioverter-defibrillator shock. JAMA. 2006 Dec 20;296(23):2839-47. doi: 10.1001/jama.296.23.2839. PMID 17179461
- [Background] Flemme I, Johansson I, Stromberg A. Living with life-saving technology - coping strategies in implantable cardioverter defibrillators recipients. J Clin Nurs. 2012 Feb;21(3-4):311-21. doi: 10.1111/j.1365-2702.2011.03847.x. Epub 2011 Sep 26. PMID 21951323
- [Background] Dougherty CM, Pyper GP, Frasz HA. Description of a nursing intervention program after an implantable cardioverter defibrillator. Heart Lung. 2004 May-Jun;33(3):183-90. doi: 10.1016/j.hrtlng.2004.01.003. PMID 15136779
- [Background] Dougherty CM, Johnston SK, Thompson EA. Reliability and validity of the self-efficacy expectations and outcome expectations after implantable cardioverter defibrillator implantation scales. Appl Nurs Res. 2007 Aug;20(3):116-24. doi: 10.1016/j.apnr.2007.04.004. PMID 17693214
- [Background] Burns JL, Serber ER, Keim S, Sears SF. Measuring patient acceptance of implantable cardiac device therapy: initial psychometric investigation of the Florida Patient Acceptance Survey. J Cardiovasc Electrophysiol. 2005 Apr;16(4):384-90. doi: 10.1046/j.1540-8167.2005.40134.x. PMID 15828880
- [Background] Brink E, Alsen P, Herlitz J, Kjellgren K, Cliffordson C. General self-efficacy and health-related quality of life after myocardial infarction. Psychol Health Med. 2012;17(3):346-55. doi: 10.1080/13548506.2011.608807. Epub 2012 Jan 31. PMID 22292865
- [Background] Barisone M, Ghirotto L, Hayter M, Molin AD, Hendriks J, Jennings C. Improving the experience of patients living with an implantable cardioverter defibrillator. Eur J Cardiovasc Nurs. 2023 Apr 12;22(3):e21-e24. doi: 10.1093/eurjcn/zvad020. No abstract available. PMID 36749003
- [Background] Baddour LM, Epstein AE, Erickson CC, Knight BP, Levison ME, Lockhart PB, Masoudi FA, Okum EJ, Wilson WR, Beerman LB, Bolger AF, Estes NA 3rd, Gewitz M, Newburger JW, Schron EB, Taubert KA; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee; Council on Cardiovascular Disease in Young; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Nursing; Council on Clinical Cardiology; Interdisciplinary Council on Quality of Care; American Heart Association. Update on cardiovascular implantable electronic device infections and their management: a scientific statement from the American Heart Association. Circulation. 2010 Jan 26;121(3):458-77. doi: 10.1161/CIRCULATIONAHA.109.192665. Epub 2010 Jan 4. PMID 20048212
- [Background] Ayyaswami V, Padmanabhan DL, Crihalmeanu T, Thelmo F, Prabhu AV, Magnani JW. Mobile health applications for atrial fibrillation: A readability and quality assessment. Int J Cardiol. 2019 Oct 15;293:288-293. doi: 10.1016/j.ijcard.2019.07.026. Epub 2019 Jul 10. PMID 31327518
- [Background] Ammannaya GKK. Implantable cardioverter defibrillators - the past, present and future. Arch Med Sci Atheroscler Dis. 2020 Jul 11;5:e163-e170. doi: 10.5114/amsad.2020.97103. eCollection 2020. PMID 32832716
- [Background] Altıkardeş ZA, Bajgora M, Sarıkaya U, Doğan B, Fak AS. Yeni bir yaklaşımla genç bireylerde kalp sağlığı takibi için web ve mobil uygulama geliştirilmesi. International Journal of Advances in Engineering and Pure Sciences. 2019;31(4):328-335.
- [Background] Al-Khatib SM, Stevenson WG, Ackerman MJ, Bryant WJ, Callans DJ, Curtis AB, Deal BJ, Dickfeld T, Field ME, Fonarow GC, Gillis AM, Granger CB, Hammill SC, Hlatky MA, Joglar JA, Kay GN, Matlock DD, Myerburg RJ, Page RL. 2017 AHA/ACC/HRS Guideline for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2018 Oct 2;72(14):e91-e220. doi: 10.1016/j.jacc.2017.10.054. Epub 2018 Aug 16. No abstract available. PMID 29097296
- [Background] Alkan H. İmplante Edilebilen Kardiyoverter Defibrilatör Hastalarında Psikososyal Faktörlerin İncelenmesi. İ.Ü. Sağlık Bilimleri Enstitüsü, Doktora Tezi, 2014, İstanbul (Danışman: Prof. Dr. Nuray Enç).
- [Background] Akay B, Oğuz S. The effect of education, telephone monitoring on self-efficacy and shock anxiety of ımplantable cardioverter defibrillator patients. Clinical and Experimental Health Sciences, 2023;13(4):855-862.
- [Background] Abbasi M, Negarandeh R, Norouzadeh R, Shojae Mogadam AR. The Challenges of Living With an Implantable Cardioverter Defibrillator: A Qualitative Study. Iran Red Crescent Med J. 2016 Jun 22;18(10):e25158. doi: 10.5812/ircmj.25158. eCollection 2016 Oct. PMID 28180011
- See also: American Heart Association (AHA). (2022a). Devices that may ınterfere with ICDs and pacemakers — https://www.heart.org/en/health-topics/arrhythmia/prevention--treatment-of-arrhythmia/devices-that-may-interfere-with-icds-and-pacemakers
- See also: American Heart Association. (AHA) (2022b). Implantable cardioverter defibrillator (ICD) — https://www.heart.org/en/health-topics/arrhythmia/prevention--treatment-of-arrhythmia/implantable-cardioverter-defibrillator-icd
- See also: American Heart Association. (AHA) (2022c). Living with your ımplantable cardioverter defibrillator (ICD) — https://www.heart.org/en/health-topics/arrhythmia/prevention--treatment-of-arrhythmia/living-with-yourimplantable-cardioverter-defibrillator-icd
- See also: NHLBI- National Heart, Lung, and Blood Institute, Defibrillators — http://www.nhlbi.nih.gov/health/dci/Diseases/icd/icd_all.html
- See also: WHO, We Are Social & Hootsuite. Digital 2022 global overwiev report. 2022 — https://wearesocial.com/uk/blog/2022/01/digital-2022-another-year-of-bumper-growth-2/2022